CLINICAL TRIAL: NCT07069036
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Food Effect of SEP-631 in Healthy Adult Volunteers
Brief Title: A Study to Evaluate Single and Multiple Doses of SEP-631 in Healthy Adult Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Septerna, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP-631-101
Record Dates: First submitted 2025-06-30; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single Ascending Dose (Experimental)
  Interventions: Drug: SEP-631; Other: Placebo
- Multiple Ascending Dose (Experimental)
  Interventions: Drug: SEP-631; Other: Placebo
- Food Effect (Experimental)
  Interventions: Drug: SEP-631

INTERVENTIONS:
Drug: SEP-631 — Oral, tablet
Other: Placebo — Oral, tablet
  Arms: Multiple Ascending Dose; Single Ascending Dose

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and food effects of oral SEP-631 in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are able and willing to provide informed consent
2. Aged 18 to 60 years at the time of consent
3. Have a BMI within the range 18.5 to 32.0 kg/m2
4. In general good health

Exclusion Criteria:

1. Any condition, which in the investigator's opinion might jeopardize participant's safety or compliance with the protocol.
2. Have a history of any severe allergic reaction or anaphylaxis
3. Have clinically significant abnormalities on clinical laboratory results.
4. Participation in other clinical trials recently/currently

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of treatment emergent adverse events | From enrollment to end of follow up visit, up to approximately 2 months

SECONDARY OUTCOMES:
Plasma PK of SEP-631 after single and multiple doses | From enrollment to end of treatment period, up to approximately 14 days
  Maximum Plasma Concentration (Cmax) of SEP-631
Plasma PK of SEP-631 under fed and fasted conditions | From enrollment to end of treatment period, up to approximately 14 days
  Maximum Plasma Concentration (Cmax) of SEP-631
Plasma PK of SEP-631 after single and multiple doses | From enrollment to end of treatment period, up to approximately 14 days
  Elimination half=life (T 1/2) of SEP-631
Plasma PK of SEP-631 after single and multiple doses | From enrollment to end of treatment period, up to approximately 14 days
  Area Under the Concentration-time Curve (AUC) of SEP-631
Plasma PK of SEP-631 under fed and fasted conditions | From enrollment to end of treatment period, up to approximately 14 days
  Area Under the Concentration-time Curve (AUC) of SEP-631